CLINICAL TRIAL: NCT02426450
Title: RFA Combined With Oxaliplatin + 5-FluoroUracil/LeucoVorin (5-FU/LV) (FOLFOX4) for Recurrent HCC:an Open Lable, Single-arm, Prospective Study
Brief Title: RFA Combined With Oxaliplatin + 5-FluoroUracil/LeucoVorin (5-FU/LV) (FOLFOX4) for Recurrent HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, M.D.,Ph.D., Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC001
Record Dates: First submitted 2015-04-16; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RFA+FOLFOX4 (Experimental): RFA:
  RFA was performed by using a commercially available system (RF 2000; Radio-Therapeutics Mountain View, CA), and a needle electrode with a 15 Ga insulated cannula with 10 hook-shaped expandable electrode tines with a diameter of 3.5 cm at expansion (LeVeen; RadioTherapeutics).
  Oxaliplatin + 5-Fluorouracil/Leucovorin:
  4 weeks after RFA; Drug: Oxaliplatin + 5-Fluorouracil/Leucovorin Day 1: Oxaliplatin 85mg/m² 2h IV infusion, leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m2 22h IV infusion.
  Day 2: Leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m² 22h IV infusion.
  Repeated every 2 weeks
  Interventions: Procedure: RFA; Drug: Oxaliplatin; Drug: 5-Fluorouracil/Leucovorin

INTERVENTIONS:
Procedure: RFA — RFA:
  RFA was performed by using a commercially available system (RF 2000; Radio-Therapeutics Mountain View, CA), and a needle electrode with a 15 Ga insulated cannula with 10 hook-shaped expandable electrode tines with a diameter of 3.5 cm at expansion (LeVeen; RadioTherapeutics).
Drug: Oxaliplatin — 4 weeks after RFA; Drug: Oxaliplatin Day 1: Oxaliplatin 85mg/m² 2h IV infusion. Repeated every 2 weeks
Drug: 5-Fluorouracil/Leucovorin — 4 weeks after RFA; Drug: 5-Fluorouracil/Leucovorin Day 1, after Oxaliplatin 85mg/m² 2h IV infusion: Leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m2 22h IV infusion.
  Day 2: Leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m² 22h IV infusion.
  Repeated every 2 weeks

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world. Partial hepatectomy and liver transplantation are considered to be standard curative therapies for HCC. When surgery is not possible, percutaneous ablation is usually considered to be alternative treatments for HCC. Recurrence is the most frequent serious adverse event observed during the follow-up of HCC patients treated for cure. Repeat hepatectomy is an effective treatment for HCC recurrence, with a 5-year survival rate of 19.4 to 56%. Unfortunately, repeat hepatectomy can be performed only in a small proportion of patients with HCC recurrence (10.4 to 31%), either because of the poor functional liver reserve or because of widespread recurrence. Radiofrequency ablation has been considered to be one of the most effective percutaneous ablations for early-stage HCC in patients with or without surgical prospects. Studies using RFA to treat HCC recurrence after hepatectomy have reported a 3-year survival rate of 62% to 68%, which is comparable to those achieved by surgery. RFA is particularly suitable to treat HCC recurrence after hepatectomy because these tumors are usually detected when they are small, and because RFA causes the least deterioration of liver function in the patients. However, according to our previous study, investigators found the recurrent rate after RFA was higher than 60%. Systemic chemotherapy is considered to be one of the main treatments for malignant tumors. HCC is known to be highly refractory to conventional systemic chemotherapy because of its heterogeneity and multiple etiologies. Before the advent of the molecular-targeted agent sorafenib, which has subsequently become the standard of care, no standard systemic drug or treatment regimen had shown an obvious survival benefit in HCC. Nowadays, there is no systemic chemotherapy regimen had been definitively recommended as the standard for treating HCC. Clinical activity of several regimens containing oxaliplatin (OXA) in advanced HCC had been demonstrated in phase II studies. In a phase II study of the FOLFOX4 (infusional fluorouracil [FU], leucovorin[LV], and OXA) regimen in Chinese patients with HCC, median overall survival (OS) was 12.4 months, mean time to progression was 2.0 months, and the response rate (RR) was 18.2%. The safety profile was acceptable. Recently, the results of a phase Ⅲ randomize study showed that FOLFOX4 served as palliative chemotherapy can induce higher overall survival, progression-free survival and response rate comparing to doxorubicin in patients with advanced hepatocellular carcinoma from Asia. The safety data was also acceptable. Therefore, investigators considered RFA to be an effective treatment for HCC recurrence after curative treatment. So our hypothesis is that RFA combined with FOLFOX4 can reduce high recurrence rate after RFA for recurrent HCC after hepatectomy. The aim of this open-lable, single prospective study is to evaluate the efficacy and safety of RFA combined with FOLFOX4 systemic chemotherapy for recurrent HCC after partial hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 75 years;
2. recurrence of HCC 12 months after initial hepatectomy;
3. no other treatment received except for the initial hepatectomy;
4. Single tumor≤5cm in diameter; or 2-3 lesions each ≤ 3.0 cm
5. lesions visible on ultrasound and with an acceptable and safe path between the lesion and the skin as shown on ultrasound;
6. no severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3;
7. Eastern Co-operative Oncology Group performance(ECOG) status 0 -1

Exclusion Criteria:

1. severe coagulation disorders (prothrombin activity <40% or a platelet count of <40,000 / mm3);
2. Child-Pugh class C liver cirrhosis or evidence of hepatic decompensation including ascites, esophageal or gastric variceal bleeding, or hepatic encephalopathy;
3. Documented allergy to platinum compound or to other study drugs; Any previous oxaliplatin or doxorubicin treatment, except adjuvant treatment more than 12 months before the randomization.
4. Previous or concurrent cancer that is distinct in primary site or histology from HCC
5. History of cardiac disease congestive heart failure > New York Heart Association (NYHA) class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted); cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin; uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
6. Active clinically serious infections (> grade 2 National Cancer Institute [NCI]- Common Terminology Criteria for Adverse Events [CTCAE] version 3.0) contraindications to carboplatin, epirubicin, mitomycin, lipiodol;
7. Pregnant or breast-feeding patients;
8. contraindications to RFA；
9. Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study;
10. Known history of human immunodeficiency virus (HIV) infection
11. Patients concomitantly receiving any other anti-cancer therapy, including interferon-α and herbal medicine which was approved by local authority to be used as "anti-cancer" medicine, except radiotherapy to non-target lesion (bone metastasis, etc)
12. Do not give written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years
Safety and Tolerability | 2 years
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

SECONDARY OUTCOMES:
Recurrence-free survival | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhen-Wei Peng, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Qin S, Bai Y, Lim HY, Thongprasert S, Chao Y, Fan J, Yang TS, Bhudhisawasdi V, Kang WK, Zhou Y, Lee JH, Sun Y. Randomized, multicenter, open-label study of oxaliplatin plus fluorouracil/leucovorin versus doxorubicin as palliative chemotherapy in patients with advanced hepatocellular carcinoma from Asia. J Clin Oncol. 2013 Oct 1;31(28):3501-8. doi: 10.1200/JCO.2012.44.5643. Epub 2013 Aug 26. PMID 23980077
- [Background] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991
- [Background] Peng ZW, Zhang YJ, Liang HH, Lin XJ, Guo RP, Chen MS. Recurrent hepatocellular carcinoma treated with sequential transcatheter arterial chemoembolization and RF ablation versus RF ablation alone: a prospective randomized trial. Radiology. 2012 Feb;262(2):689-700. doi: 10.1148/radiol.11110637. Epub 2011 Dec 12. PMID 22157201